CLINICAL TRIAL: NCT00956904
Title: Ultrasound-Guided Navigation in Robot-Assisted Laparoscopic Radical Prostatectomy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: IRB approval expired.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Misop Han, Associate Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00027540
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostatectomy; Transrectal Ultrasound; Tandem RALP
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3-D TRUS navigation software during T-RALP (Experimental)
  Interventions: Device: 3-D TRUS navigation software during T-RALP

INTERVENTIONS:
Device: 3-D TRUS navigation software during T-RALP — A new solution for guiding the surgeon in RALP is image-guided navigation using transrectal ultrasound (TRUS). A TRUS-guided intraoperative navigation system using a robotic ultrasound probe manipulator (TRUS Robot) has been developed. The research is a pilot clinical trial of the TRUS Robot and three-dimensional (3-D) navigation software to test its image-guidance ability of helping the surgeon during RALP. This is a dual robot approach, a Tandem-RALP (T-RALP). The TRUS Robot allows a steady holding as well as remote manipulation of the TRUS probe. In addition, the TRUS Robot can track the accurate position of TRUS probe which allows 3-D reconstruction of the images.

SUMMARY:
A new solution for guiding the surgeon in robot-assisted laparoscopic radical prostatectomy (RALP) is image-guided navigation using transrectal ultrasound (TRUS). A TRUS-guided intraoperative navigation system using a robotic ultrasound probe manipulator (TRUS Robot) has been developed. The proposed research is a pilot clinical trial of the TRUS Robot and three-dimensional (3-D) navigation software to test its image-guidance ability of helping the surgeon during RALP. This is a dual robot approach, a Tandem-RALP (T-RALP). The TRUS Robot allows a steady holding as well as remote manipulation of the TRUS probe. In addition, the TRUS Robot can track the accurate position of TRUS probe which allows 3-D reconstruction of the images. While the intraoperative TRUS findings will not be used in surgical decision making in this trial, the use of TRUS imaging during radical prostatectomy can potentially improve the visualization of the NVB and subsequently improve postoperative recovery of potency in men. In addition, the 3-D reconstruction images of the prostate gland can potentially provide clear and accurate guidance of surgical landmarks to the surgeon..

DETAILED DESCRIPTION:
The preservation of the neurovascular bundle (NVB) including cavernous nerves during radical prostatectomy improves the postoperative recovery of sexual potency. At present, the location of NVB is determined by the surgeon's visual estimation. However, NVB is difficult to visualize with simple visual magnification of the surgical field with surgical loupes or laparoscopic lenses due to the periprostatic connective tissue and intraoperative hemorrhage. One approach to better estimate the location of the NVB is to identify a macroscopic landmark to more clearly direct the surgeon to the location of the NVB. The accompanying arteries and veins in the NVB, which are visible with Doppler ultrasound, can serve as a macroscopic landmark to localize the microscopic cavernous nerves in the NVB. Therefore, the use of TRUS imaging during radical prostatectomy can potentially improve the visualization of the NVB and subsequently improve postoperative recovery of potency in men. In addition, the 3-D shape of the prostate gland can potentially be clearly and accurately delineated in ultrasounds imaging, providing direct guidance of landmarks to the surgeon.

Recently, intraoperative TRUS imaging has been used to visualize the prostate gland and NVB during laparoscopic radical prostatectomy (LRP). The investigators reported that the intraoperative use of TRUS was helpful in imaging the location and local extent of hypoechoic area(s), providing real-time guidance for the surgeon during NVB release and apical dissection of the prostate, and monitoring a calibrated, lobe-specific, wider dissection around a cancer nodule with suspected extracapsular extension (ECE). With the enhanced visualization of the surgical field by TRUS imaging, they reported significant improvement in NVB preservation and a decreasing rate of positive surgical margin, which is a surrogate for the technical quality of the surgery. However, several aspects related most likely to technology limitations can further be improved. For example, the TRUS probe was manipulated by a human assistant during LRP, compromising image stability especially with Doppler imaging, discarding the pose of the images, and performing navigation based on the recommendations of the assistant rather than using an actual navigation software. Moreover, their application of TRUS can be used in the non-robotic LRP only, because the daVinci® robot used in RALP occupies the place of a human assistant at the end of the operative table. Finally, there was no objective measure to quantify the performance of the navigational aid.

Regardless of the study's shortcomings, the authors reported that their positive surgical margin rates decreased precipitously since their use of the TRUS guidance, demonstrating potential benefit of the TRUS-based guidance during surgery. Since their study, the use of intraoperative TRUS guidance during prostate surgery has not gained wide acceptance, and was, in fact, criticized because it requires an additional personnel with an expertise in TRUS. Alternatively, we propose to use the TRUS Robot, a robotic arm to hold and manipulate the TRUS probe remotely, allowing the surgeon to manipulate the TRUS probe without the need for a human assistant during RALP. We also propose to use 3-D TRUS navigation with the images obtained by the TRUS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be scheduled for a robotic LRP
* Patients must be between the ages of 35 and 75
* Patients must not have one of the listed exclusion criteria
* Patients must be able to understand and willing to adhere to the study protocol
* Patients must have a clinical stage diagnosis of T1 or T2
* Patients must have a preoperative serum PSA < 20ng/ml
* Patients must have a biopsy Gleason score of 5-8

Exclusion Criteria:

* Patients less than 35 years of age and over 75 years of age.
* Patients with previous rectal surgery
* Patients with anal stenosis that prevents the TRUS probe insertion
* Patients with extensive abdominal surgery
* Patients with inadequate bowel prep
* Patients who are unwilling or unable to sign informed consent
* Patients on anticoagulation medication (eg. coumadin, lovenox, or heparin)
* Patients with a clinical stage diagnosis of T3 - Patients with a preoperative serum PSA ≥ 20 ng/mL
* Patients with a biopsy Gleason score < 5 or > 8

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of TRUS Robot and 3-D TRUS navigation software. | Measurements will be recorded in the time frame between the start of surgery to the end of surgery.
  To assess whether NVB localization is accurate using the TRUS Robot and 3-D TRUS navigation software during T-RALP & can accurately locate and quantify the distance between anatomical landmarks.

SECONDARY OUTCOMES:
Safety of T-RALP | Measurements determined by Dr. Han will be recorded in the time frame between the start of surgery to the end of surgery.
  To determine T-RALP can be safely performed without increased complications including rectal injury.

CONTACTS AND LOCATIONS:
Overall Officials: Misop Han, M.D., M.S., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States